CLINICAL TRIAL: NCT03696537
Title: A Dose Escalation Study of Intensity Modulated Total Marrow Irradiation (IMRT-TMI) With Fludarabine as a Myeloablative Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Relapsed and Refractory Hematologic Malignancies
Brief Title: IMRT-TMI With Fludarabine as Myeloablative Conditioning for Allogeneic HSCT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Extreme toxicity
Sponsor: Naoyuki G. Saito, M.D., Ph.D. (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor-Investigator, Naoyuki G. Saito, M.D., Ph.D., Assistant Professor of Radiation Oncology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0652
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Acute Myeloid Leukemia; Chronic Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndromes
Keywords: Radiation; Total Marrow Irradiation; Fludarabine; Bone Marrow Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — fludarabine

STUDY DESIGN:
Intervention Model Description: Standard "3+3" phase I design of dose escalation using 3 patients per dose level cohort with an expansion to 6 patients at the MTD will be used in Phase I. We will treat 3 patients at the initial dose level of TMI. If no dose-limiting toxicity (DLT) is observed, the next cohort of three patients is treated at the next higher dose level. If 1 of the 3 patients demonstrates DLT, an additional 3 patients are treated at that dose level. If only 1 of the 6 shows DLT, the next cohort of three patients is entered at the next dose level. If 2 or more of the 6 demonstrate DLT, the MTD is defined as the previous dose level. If no DLT is observed in the final dose level, the number of patients treated will be expanded to 6. In phase II, we will enroll additional patients at the defined MTD level.
  *Stopping criteria was met during the first dose level cohort in Phase l. The trial will not continue into Phase II as originally planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Total Marrow Irradiation (Experimental)
  Interventions: Drug: Fludarabine; Radiation: Total Marrow Irradiation (TMI)

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2/day IV (total 5 doses) administered days -7 through -3 of conditioning regimen
Radiation: Total Marrow Irradiation (TMI) — TMI will be delivered twice a day, at least 6 hours apart, on days -7 through -3 (total of 10 fractions) of conditioning regimen

SUMMARY:
This is a phase I/II clinical trial on the use of total marrow irradiation (TMI) given concurrently with fludarabine, a chemotherapy drug commonly used to treat leukemia, as a myeloablative therapy for patients undergoing Allo-HSCT. TMI is a targeted technique to deliver radiation to the bone marrow while minimizing dose to other normal organs in the body. In phase I of the clinical study, the dose of radiation to the bone marrow will be incrementally increased to determine the highest tolerated TMI dose. In phase II, the effectiveness of the TMI-fludarabine conditioning regimen utilizing that dose of radiation will be studied. Acute and long-term toxicity data as well as quality of life data will also be studied.

*Stopping criteria was met during the first dose level cohort in Phase l. The trial will not continue into Phase II as originally planned.

DETAILED DESCRIPTION:
This is a phase I/II clinical trial to determine the maximum tolerated dose (MTD) of intensity modulated radiation therapy based total marrow irradiation (TMI) concurrent with fludarabine as a myeloablative conditioning regimen for allogeneic hematopoietic stem cell transplantation (Allo-HSCT), as well as to determine the efficacy of the regimen in patients with high-risk and relapsed or refractory leukemia and myelodysplasia. TMI, which allows for conformal dosing of target bone marrow tissue while giving lower doses to organs at risk, is considered by many to be a superior alternative to conventional total body irradiation (TBI)

Primary Objectives:

Phase I:

Determine the MTD of TMI given concurrently with fludarabine (fixed at 150 mg/m2) as a conditioning regimen for Allo-HSCT for patients with high risk (relapsed/refractory) acute lymphocytic leukemia (ALL), acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), and chronic myelogenous leukemia (CML).

Phase II:

Single-arm exploratory study to expand the cohort at the MTD level to estimate 1- year overall survival (OS), with the objective of increasing the OS from the historical rate of 30% (null hypothesis ) to 50% (alternate hypothesis) with 80% power and a one-sided type I error of 0.05.

Secondary Objectives

1. Describe the extramedullary toxicity and the incidence of complications, including mucositis, acute and chronic graft versus host disease (GvHD), sinusoidal obstruction syndrome (SOS), and pneumonitis.
2. Describe the time to engraftment of neutrophils and platelets
3. Describe the disease response rate at day 30 after transplantation
4. Describe the overall survival and disease-free survival
5. Describe the cumulative incidence of relapse and non-relapse mortality
6. Determine the correlation between plasma/serum markers and radiation induced acute and long term toxicities.
7. Describe the quality of life metrics of participating subjects

   * Stopping criteria was met during the first dose level cohort in Phase l. The trial will not continue into Phase II as originally planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with one of the following conditions:

   Acute Myeloid Leukemia (AML) who are not in complete remission, and who have either primary refractory or relapsed disease, and who do not have more than one of the following adverse factors:
   1. Duration of first CR < 6 months (if previously in CR)
   2. Poor risk karyotype including any of the following: complex karyotype with ≥3 clonal abnormalities, 5q-/-5, 7q-/-7, 11q23 abnormalities, inv(3q), 20q or 21q abnormalities, t(6;9), t(9;22), 17p abnormalities [or TP53 mutations] or monosomal karyotype. Molecular typing (except for TP53 mutation) will not be used for eligibility criteria determination.
   3. Circulating peripheral blood blasts at time of enrollment
   4. Karnofsky performance status <90%

   Acute Lymphocytic Leukemia (ALL) who are not in complete remission, and who have either primary refractory or relapsed disease, and who do not have more than one of the following adverse factors:
   1. First refractory relapse. Patients in second or subsequent relapse are excluded.
   2. Donor is CMV seropositive
   3. Bone marrow blasts >25% (within 30 days of admission)
   4. Age >40 years

   Myelodysplasia with a Revised International Prognostic Score (IPSS-R) of greater than 4.5 (i.e., high- or very-high risk).

   Chronic Myelogenous Leukemia (CML) in either
   1. Accelerated phase, defined by any of the following:

      * 10-19% blasts in peripheral blood white cells or bone marrow
      * Peripheral blood basophils at least 20%
      * Persistent thrombocytopenia (<100 x 109/l) unrelated to therapy, or persistent thrombocytosis (>1000 x 109/l) unresponsive to therapy
      * Increasing spleen size and increasing white blood cell (WBC) count unresponsive to therapy
      * Cytogenetic evidence of clonal evolution (i.e., the appearance of an additional genetic abnormality that was not present in the initial specimen at the time of diagnosis of chronic phase)
   2. Chronic phase provided a complete hematologic remission was not achieved by 3 months or a complete cytogenetic remission by 18 months and the patient had received at least 2 tyrosine kinase inhibitors.
2. Patient age 18-65 years old at time of consent
3. Availability of a consenting human leukocyte antigens(HLA) -matched donor
4. Karnofsky Performance Status 70% or higher
5. Required baseline laboratory values:

   1. Estimated creatinine clearance ≥ 60 ml/min
   2. Aspartate aminotransferase and alanine aminotransferease ≤ 2.5 x upper limit of normal value
   3. Bilirubin ≤ 1.5 x upper limit of normal value
6. Required baseline cardiac function of left ventricular ejection fraction (LVEF) > 45

   * corrected
7. Required baseline pulmonary function of lung diffusing capacity (DLCO) > 45 % predicted (corrected for hemoglobin)
8. Patient must be capable of understanding the investigational nature of this study, potential risks and benefits of the study, and be able to provide a valid informed consent.

Exclusion Criteria:

1. Patients with ALL who are in second or subsequent relapse
2. HIV seropositive patients.
3. Pregnant or nursing females are excluded from this study.
4. Prior radiation therapy
5. Patients who have had a prior autologous or allogeneic bone marrow or stem cell transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of Total Marrow Irradiation (TMI) in combination with 150 mg/m2 fludarabine- Phase I only | Day -7 of conditioning regimen through 30 days post transplant (37 days)
Maximum-tolerated dose (MTD) of Total Marrow Irradiation (TMI) in combination with 150 mg/m2 fludarabine-Phase I only | Day -7 of conditioning regimen through 30 days post transplant (37 days)
Overall survival (OS) rate 1 year post transplant-Phase II only | 1 year

SECONDARY OUTCOMES:
Frequency of non hematologic toxicities | 100 days
Incidence of infection | 100 days
Type of infections | 100 days
Incidence of graft versus host disease (GvHD) | 100 days
Incidence of chronic graft versus host disease (GvHD) | 2 years
Incidence of sinusoidal obstruction syndrome (SOS) | 100 days
Incidence of pneumonitis | 100 days
Incidence of mucositis | 100 days
Time to engraftment of neutrophils | from date of transplant to the first of three consecutive days after transplantation during which the absolute neutrophil count (ANC) is greater than or equal to 0.5 x 10^9/liter
Time to engraftment of platelets | from date of transplant until he first of seven consecutive days after transplantation during which the platelet count is greater than or equal to 20 x10^9/liters without transfusion.
Disease response rate | Day 30 after transplant (30 days)
Incidence of relapse mortality | 30 days
Incidence of relapse mortality | 100 days
Incidence of relapse mortality | 1 year
Incidence of non-relapse mortality | 30 days
Incidence of non-relapse mortality | 100 days
Incidence of non-relapse mortality | 1 year
Disease-Free Survival | 2 years
Mean Quality of Life (QOL) as measured by Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) version 4 | Screening (at simulation), day +180, day +365, + 2 years from transplant (approximately 2 years)
  50 item likert type scale with responses measuring from 0-4 (where 0 = not at all; 1 = a little bit; 2 = somewhat, 3 = quite; and 4 = very much) with higher scores correlating to higher QOL

CONTACTS AND LOCATIONS:
Overall Officials: Naoyuki G Saito, MD PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States